CLINICAL TRIAL: NCT04876885
Title: The Future of Viral Communications: Video-Based Health Promotion Strategies for COVID-19 Vaccinations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Sarrah Lal, Assistant Professor, McMaster University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12902
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Health Promotion; Health Education; COVID-19 Vaccines
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: This study looks at two groups. First, it directly measures response of COVID-19 vaccine hesitancy in the general public to education videos on COVID-19 vaccine development, validation, and dissemination. Second, it surveys two stakeholder groups - healthcare professionals and public health professionals to better understand their evaluation of COVID-19 vaccine education needs in the general public, based on their interpretation of commonly asked questions, best practices in health promotion, and evaluation of information already available.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General public (Other): The individuals recruited to the study will include those who are age 16 and older. Due to recruitment feasibility we will focus efforts on individuals living in Ontario. We intend to recruit individuals from COVID-19 assessment centres that are partnering in our study as well as through social media posts (Facebook, Twitter, LinkedIn).
  Interventions: Other: Educational video
- Healthcare professionals and public health professionals (Other): The individuals recruited to the study will include healthcare professionals and public health professionals impacted by infectious disease outbreaks. Social media will be used to disseminate surveys to physicians, nurses, nurse practitioners, pharmacists, and healthcare workers. Public health units will disseminate surveys to their workforce.
  Interventions: Other: Educational video

INTERVENTIONS:
Other: Educational video — Three two-minute educational videos about COVID-19 vaccine development and dissemination

SUMMARY:
The investigators aim to study whether education, in the form of three two-minute educational videos about COVID-19 vaccine development and dissemination, reduces vaccine hesitancy and increases intent to vaccinate. The investigators intend to use insights from this research study to develop a framework for video-based 'education prescriptions' that reduce vaccine hesitancy and increase intent to vaccinate across a number of infectious diseases. This may have wide-ranging impact: inform practice for health promotions and public health, as well as support infectious disease related work done by healthcare professionals (e.g. those working in travel medicine, where vaccination rates are also low).

DETAILED DESCRIPTION:
The World Health Organization listed vaccine hesitancy as one of the leading threats to global health in 2019. Vaccine hesitancy is defined as the "reluctance or refusal to vaccinate despite the availability of vaccines". Given the novelty of the COVID-19 pandemic, hesitancy towards use of COVID-19 vaccine may be linked to the process of vaccine development and clinical trial validation of safety and/or efficacy, rather than hesitations regarding vaccines in general. This has already inspired several education campaigns. It is unclear whether education leads to reduced hesitance and whether reduced hesitance leads to increased intent to vaccinate. Further, early surveys demonstrating high COVID-19 vaccine acceptance and intent to vaccinate may not reflect actual uptake, as shown by comparisons to flu vaccination uptake at a time when flu vaccines are both available, validated and largely freely accessible. Inspiring vaccine confidence is a multifaceted challenge, and the COVID-19 pandemic has shed light on one of its aspects, specifically the public health approach to health information dissemination. The lack of evidence-based knowledge and preparedness coupled with pandemic fatigue impacts the uptake of recommended health behaviours and puts human lives at risk. Different people adopt different responses to health promotion materials based on a variety of socioeconomic factors. For example, in an American study on vaccination in children, it was found that children who had never received a vaccine tended to come from affluent, college educated families, while those who had only received some recommended vaccinations came from minority families that were single parent, low-income and less likely to have completed higher education. Almost 50% of the parents of the unvaccinated children cited concerns about vaccine safety. The strength of beliefs leading to hesitancy may change the ability to affect intent to vaccinate. These beliefs may be contributed to by cultural dimensions in Canada and cultures of recently immigrated individuals, with regards to individualism, collectivism, perceptions of social benefits, etc. These factors might also impact the choice to vaccinate. The existence of many outlets for highly varied information underscores the need for unbiased and credible education on COVID-19 vaccinations. The investigators aim to study whether education, in the form of three two-minute educational videos about COVID-19 vaccine development and dissemination, reduces vaccine hesitancy and increases intent to vaccinate. The investigators intend to use insights from this research study to develop a framework for video-based 'education prescriptions' that reduce vaccine hesitancy and increase intent to vaccinate across a number of infectious diseases. This may have wide-ranging impact: inform practice for health promotions and public health, as well as support infectious disease related work done by healthcare professionals (e.g. those working in travel medicine, where vaccination rates are also low).

ELIGIBILITY:
Inclusion Criteria:

For the general public arm:

* An understanding of the English language at a grade 8 written level
* Reside in Ontario

For the healthcare professionals and public health professionals arm:

* Licensed to practice as a healthcare professional in Ontario
* An understanding of the English language at a grade 8 written level
* Reside in Ontario

Exclusion Criteria:

* Any individuals under age 16

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-06 (Estimated); Primary Completion 2021-06-06 (Estimated); Study Completion 2021-06-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants indicating intent to vaccinate against COVID-19 | One month
  The primary end point of the study is "intent to vaccinate against COVID-19" within the general public survey. We are looking for an increase in intent to vaccinate after the educational videos are completed. This is a yes/no answer choice. A change in response may be indicative of the impact of education on vaccination intent.

SECONDARY OUTCOMES:
Change in score regarding vaccine hesitation after exposure to educational materials | One month
  The study seeks to understand whether providing video-based educational materials yields a positive change in score regarding vaccine hesitation (at least one point decrease) after exposure to educational materials. A change in score may indicate that educational materials support a decrease in COVID-19 vaccination hesitancy in the population. The scale title will be "Level of concern about the COVID-19 vaccine". Values will range from 1-5, where 1 indicates no concern and 5 indicates high concern.

CONTACTS AND LOCATIONS:
Overall Officials: Sarrah M Lal, MBA, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malik AA, McFadden SM, Elharake J, Omer SB. Determinants of COVID-19 vaccine acceptance in the US. EClinicalMedicine. 2020 Sep;26:100495. doi: 10.1016/j.eclinm.2020.100495. Epub 2020 Aug 12. PMID 32838242
- [Background] Harrison EA, Wu JW. Vaccine confidence in the time of COVID-19. Eur J Epidemiol. 2020 Apr;35(4):325-330. doi: 10.1007/s10654-020-00634-3. Epub 2020 Apr 22. PMID 32318915
- [Background] Dodd RH, Cvejic E, Bonner C, Pickles K, McCaffery KJ; Sydney Health Literacy Lab COVID-19 group. Willingness to vaccinate against COVID-19 in Australia. Lancet Infect Dis. 2021 Mar;21(3):318-319. doi: 10.1016/S1473-3099(20)30559-4. Epub 2020 Jun 30. No abstract available. PMID 32619436
- [Background] Edwards B, Biddle N, Gray M, Sollis K. COVID-19 vaccine hesitancy and resistance: Correlates in a nationally representative longitudinal survey of the Australian population. PLoS One. 2021 Mar 24;16(3):e0248892. doi: 10.1371/journal.pone.0248892. eCollection 2021. PMID 33760836
- [Background] Sherman SM, Smith LE, Sim J, Amlot R, Cutts M, Dasch H, Rubin GJ, Sevdalis N. COVID-19 vaccination intention in the UK: results from the COVID-19 vaccination acceptability study (CoVAccS), a nationally representative cross-sectional survey. Hum Vaccin Immunother. 2021 Jun 3;17(6):1612-1621. doi: 10.1080/21645515.2020.1846397. Epub 2020 Nov 26. PMID 33242386
- See also: Importance of targeted messaging in getting people to adhere to COVID-19 safety measures — https://www.concordia.ca/news/stories/2020/09/15/global-covid-19-study-finds-a-strong-link-between-health-messaging-and-behaviour.html